CLINICAL TRIAL: NCT07098637
Title: The Effect of a Self-Compassionate Mindfulness Psychoeducation Program Implemented in Prison on Internalized Stigma, Emotion Regulation, and Forgiveness in Juvenile Delinquents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Abdullah Usta, lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2024-142
Record Dates: First submitted 2025-07-23; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Juvenile Delinquency
Keywords: Self-Compassion; Forgiveness; Stigmatization; Emotion Regulation; juvenile delinquency
MeSH Terms: conditions — Stereotyping; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: To prevent bias and enhance internal validity, the processes of randomization and blinding were structured in accordance with the physical layout of the correctional facility. The institution consists of two separate blocks (Block A and Block B), and this architectural structure served as the basis for implementing randomization. A total of 68 delinquent adolescents who met the inclusion criteria were assigned to experimental and control groups using block-based simple randomization. Accordingly, 34 participants from Block A were randomly assigned to the experimental group, and 34 participants from Block B were randomly assigned to the control group, ensuring an unbiased distribution. Placement into blocks was conducted without regard to individual characteristics, and equal block capacity was considered to ensure intra-block homogeneity. This approach enabled physical separation between the groups, preventing direct contact and facilitating effective blinding between experimental and
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): A total of 68 delinquent adolescents who met the inclusion criteria were assigned to the experimental and control groups using a block-based simple randomization method. Accordingly, 34 participants from Block A were randomly assigned to the experimental group, while 34 participants from Block B were randomly assigned to the control group in an unbiased manner. Placement into blocks was conducted without considering individual characteristics, and equal capacity between blocks was ensured to maintain intra-block homogeneity. This method prevented direct interaction between groups, ensuring both physical separation and effective blinding between the experimental and control groups. Thus, participants were unaware of each other's group assignments, preserving the integrity and methodological validity of the study.
- experimental group (Experimental): A total of 68 delinquent adolescents who met the inclusion criteria were assigned to the experimental and control groups using a block-based simple randomization method. Accordingly, 34 participants from Block A were randomly assigned to the experimental group, while 34 participants from Block B were randomly assigned to the control group in an unbiased manner. Placement into blocks was conducted without considering individual characteristics, and equal capacity between blocks was ensured to maintain intra-block homogeneity. This method prevented direct interaction between groups, ensuring both physical separation and effective blinding between the experimental and control groups. Thus, participants were unaware of each other's group assignments, preserving the integrity and methodological validity of the study.
  Interventions: Behavioral: Self-Compassionate Mindfulness Psychoeducation Program

INTERVENTIONS:
Behavioral: Self-Compassionate Mindfulness Psychoeducation Program — The researcher completed the internationally accredited institutional and practical training program titled "All About Compassion in 12 Weeks: A Thousand Faces of Compassion", offered by the School of Compassion. Expert opinions were sought from the planning phase of the study for the content of the program, which was designed by the researchers. In developing the content of the Self-Compassionate Mindfulness Psychoeducation Program for Delinquent Adolescents, the opinions of three academic faculty members were consulted. Based on the suggestions received, the session titles of the psychoeducation program were determined as follows:
  1. Holding Our Own Hand: Discovering Self-Compassion
  2. Discovering Awareness of Thought
  3. Understanding Pain, Approaching with Compassion
  4. Facing Reality: Acceptance
  5. Calm Waters: Forgiveness
  6. Moving Forward, Farewell, and a New Beginning.
  Arms: experimental group

SUMMARY:
The aim of this study is to determine the effect of the Self-Compassionate Mindfulness Psychoeducation Program on internalized stigma, emotion regulation, and forgiveness among adolescents involved in delinquency under prison conditions.

Objectives

Objective 1: To develop a Self-Compassionate Mindfulness Psychoeducation Program for juveniles involved in delinquency and to ensure its content validity.

Objective 2: To conduct a pilot implementation of the developed psychoeducation program.

Objective 3: To administer pre-tests to juveniles involved in delinquency using psychometrically validated and reliable scales to assess levels of internalized stigma, emotion regulation, and forgiveness.

Objective 4: To implement the developed psychoeducation program in a prison setting over the course of six sessions.

Objective 5: To administer post-tests to juveniles involved in delinquency using psychometrically validated and reliable scales to assess levels of internalized stigma, emotion regulation, and forgiveness.

Objective 6: To perform statistical analyses of the collected data.

H₀ Hypothesis:

The Self-Compassionate Mindfulness Psychoeducation Program administered to juveniles involved in delinquency in a prison setting does not affect the mean scores of internalized stigma, emotion regulation, and forgiveness in the experimental group.

H₁a Hypothesis:

The Self-Compassionate Mindfulness Psychoeducation Program administered to juveniles involved in delinquency in a prison setting decreases the mean scores of internalized stigma in the experimental group.

H₁b Hypothesis:

The Self-Compassionate Mindfulness Psychoeducation Program administered to juveniles involved in delinquency in a prison setting increases the mean scores of emotion regulation in the experimental group.

H₁c Hypothesis:

The Self-Compassionate Mindfulness Psychoeducation Program administered to juveniles involved in delinquency in a prison setting increases the mean scores of forgiveness in the experimental group.

DETAILED DESCRIPTION:
1. Type of the Study This study was conducted using a single-blind, randomized controlled experimental design.
2. Location and Time of the Study This study was carried out between March 2025 and May 2025 with adolescents in solitary confinement who had been driven to delinquency, in the Kavak Juvenile and Youth Closed Penal Institution located in Kavak district, Samsun province. The institution consists of two separate units, Block A and Block B, with a total capacity of 350 individuals and accepted its first inmates in 2022. The Kavak Juvenile and Youth Closed Penal Institution holds the distinction of being the first and only juvenile and youth closed penal facility in the Black Sea Region.

   The self-compassionate mindfulness psychoeducation program was conducted in the group workroom located within the institution.
3. Study Population and Sample The population of the study consisted of adolescents in solitary confinement in the aforementioned penal institution, while the sample was composed of individuals meeting the study inclusion criteria. The sample size was calculated using the G*Power 3.1 program. For the variable of internalized stigma, mean scores were taken as 106.67±29.48 (group 1) and 90.00±16.91 (group 2). Based on these values, with a 95% confidence interval, 5% margin of error, 0.98 effect size, and 95% power, the required sample size was calculated to be 56.

   For the variable of emotion regulation, mean scores were 2.25±0.78 (measurement-1) and 1.91±0.75 (measurement-2) . With the same confidence interval and error rate, but a 0.45 effect size and 90% power, the required sample size was calculated as 54.

   For the forgiveness variable, mean scores were 57.92±13.34 (group-1) and 48.95±9.37 (group-2) , with a 0.78 effect size and 85% power, yielding a required sample size of 62.

   Based on these calculations, the target sample size was determined as 62 participants (31 in the experimental group and 31 in the control group). Considering possible dropouts, the study aimed to include 68 participants (34 in each group), including approximately 10% as reserves.

   Adolescents who met the inclusion criteria were assigned to the experimental or control groups based on the institution's physical layout. Participants in Block A were randomly assigned to the experimental group, and those in Block B were randomly assigned to the control group using a simple randomization method.

   The psychoeducation program for the experimental group was conducted weekly in three separate group sessions at different time slots. Each session was limited to a maximum of 11-12 participants, and groups were planned in a way to ensure that they would not see each other.

   Inclusion Criteria

   Literacy

   Ability to speak and understand Turkish

   Aged between 12 and 18

   Convicted and currently incarcerated

   Willingness to participate in the study

   Exclusion Criteria

   Unwillingness to participate

   Diagnosed with a psychiatric disorder that may disrupt group dynamics

   Younger than 12 or older than 18

   Having a physical disability that may affect participation (e.g., hearing or speech impairment)

   Withdrawal Criteria

   Requesting to withdraw during the study

   Not participating in at least one of the pre- or post-tests

   Failure to attend all sessions

   Ending of solitary confinement before the study concludes
4. Randomization and Blinding To prevent bias and increase internal validity, the processes of randomization and blinding were structured based on the institution's physical layout. The institution comprises two blocks (A and B), which were used as the basis for randomization. A total of 68 eligible adolescents were randomly assigned to experimental and control groups based on their blocks. From Block A, 34 participants were randomly selected for the experimental group, and from Block B, 34 were selected for the control group using simple randomization.

   Block assignments were made without considering individual characteristics, and capacity equality between blocks was ensured for homogeneity. The physical separation of the blocks enabled effective blinding, preventing direct contact between the groups and ensuring participants were unaware of each other's group affiliation.

   Data collected were coded as Group A and Group B and entered into SPSS. An independent statistician analyzed the coded data. After the analysis and reporting were completed, group codes were revealed. Thus, selection bias, statistical bias, and detection bias were controlled.
5. Variables of the Study Dependent Variables

   Level of Internalized Stigma

   Level of Emotion Regulation

   Level of Forgiveness

   Independent Variable

   Self-Compassionate Mindfulness Psychoeducation Program

   Control Variables

   Age

   Type of Offense
6. Data Collection Tools Data were collected using the "Adolescent Demographic Information Form," "Emotion Regulation Scale for Children and Adolescents," "Forgiveness Scale for Adolescents," and the "Internalized Stigma Scale for Children and Adolescents."

   6.1. Adolescent Demographic Information Form This form was developed based on the literature and includes questions about age and type of offense .

   6.2. Emotion Regulation Scale for Children and Adolescents

   Developed by Phillips and Power 2007 and validated in Turkish by Yıldız and Duy 2014. It consists of 18 items rated on a 5-point Likert scale and has four subscales:

   Internal Functional Emotion Regulation (IFER)

   External Functional Emotion Regulation (EFER)

   Internal Dysfunctional Emotion Regulation (IDER)

   External Dysfunctional Emotion Regulation (EDER) Higher scores indicate more frequent use of the respective regulation strategy. Test-retest reliability coefficients range between 0.51 and 0.70.

   6.3. Forgiveness Scale for Adolescents Developed by Asıcı and Karaca 2018, this 21-item, 5-point Likert scale measures adolescents' tendency to forgive in interpersonal relationships. It includes four subscales: revenge, holding onto anger, and empathy. Higher scores indicate a greater tendency to forgive. The total score ranges from 21 to 105, and the scale's Cronbach's alpha was reported as .90.

   6.4. Internalized Stigma Scale for Children and Adolescents

   Developed by Çağlayan 2019, this 32-item scale consists of six factors:

   Behavioral Problems

   Social and Academic Adjustment

   Concealing the Diagnosis

   Feelings of Exclusion

   Chronicity of the Problem

   Emotional Difficulties Items are rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).

   Reliability coefficients: Cronbach's alpha = .91 (self-perception section), .92 (perceived by others); split-half reliability = .85 and .89, respectively.
7. Designing the Self-Compassionate Awareness Psychoeducation Program for Juvenile Offenders The project coordinator has completed the institutional and practical training program titled "All About Compassion: A Thousand Faces of Compassion - 12-Week Program" from the internationally accredited School of Compassion institution. Expert opinions were obtained from the planning stage of the study for the program, the content of which was designed by the researchers. In the content planning of the Self-Compassionate Awareness Psychoeducation Program for Juvenile Offenders, the expert opinions of three faculty members were consulted. Based on the recommendations received, the session titles of the psychoeducation program were determined in sequence.
8. Pilot Study Phase A pilot study will be conducted prior to the main research in order to evaluate the strengths and areas needing improvement of the intervention. Five juvenile individuals who meet the inclusion criteria of the study will be included in this pilot study. However, these adolescents will not be included in the sample group in which the main study will be conducted.
9. Reaching the Target Group Juvenile offenders in solitary confinement at the Samsun Kavak Juvenile and Youth Closed Penal Institution will be informed about the study. The inclusion, exclusion, and withdrawal criteria for the study will be explained to the juvenile offenders. Consent will be obtained from the adolescents who volunteer to participate in the study. This process will continue until a total of 68 juvenile individuals are reached.
10. Collection of Pre-Test Data

    10.1.Pre-Test Implementation Process: Juvenile offenders who meet the inclusion criteria and are informed about the study will be included in the sample pool. In the next stage, the sample group will be divided into experimental and control groups using the Research Randomizer program.

    10.2.Randomization and Blinding Stage: To prevent bias during the research process, randomization will be concealed, and randomized assignment will be performed. A statistics expert, who is not familiar with the characteristics of the 68 juvenile offenders meeting the inclusion criteria, will carry out simple randomization to assign the participants impartially to the groups (experimental and control). As a result, 34 adolescents will be assigned to the experimental group and 34 adolescents to the control group. Until the implementation of the Self-Compassionate Awareness Psychoeducation Program begins, the group assignments of the adolescents in the experimental and control groups will be kept confidential, ensuring participant blinding. The juvenile offenders will not be aware of whether they belong to the experimental or control group. Additionally, during the data evaluation process, the data from the experimental and control groups will be coded to ensure the blinding of the statistics expert as well.

    Pre-test measurements will be administered to the juvenile offenders who are randomly assigned to the experimental and control groups through randomization. Before the implementation of the planned program, pre-test measurements will be conducted with individuals in both the experimental and control groups using the "Adolescent Descriptive Characteristics Form," "Emotion Regulation Scale for Children and Adolescents," "Forgiveness Scale for Adolescents," and the "Internalized Stigma Scale for Children and Adolescents" through the face-to-face interview technique.

    To ensure that the randomization is not compromised due to participants dropping out of the sample after randomization, the intention-to-treat (ITT) analysis will be used during the data collection process.
11. Data Collection Phase The juvenile offenders who have completed the pre-tests and are in the experimental group will be contacted, and suitable dates/times for the sessions will be determined through collaboration between the researcher and the institution. The group sessions for the juvenile offenders in the experimental group will be conducted with three experimental groups consisting of 11, 11, and 12 participants, respectively. For each of the three experimental groups, one session per week will be held, and the Self-Compassionate Awareness Psychoeducation Program, consisting of a total of 6 sessions, will be implemented face-to-face at the institution.A preparatory session was held during which the purpose, procedures, and duration of the study were explained to participants, and informed consent was obtained. Data were collected in two stages (pre-test and post-test) between March 2025 and May 2025 from the experimental group.

In the preparatory session, participants completed the pre-test instruments: "Adolescent Demographic Information Form," "Emotion Regulation Scale for Children and Adolescents," "Forgiveness Scale for Adolescents," and "Internalized Stigma Scale for Children and Adolescents." In addition, a general plan for subsequent psychoeducation sessions was created. One day before each session, the researcher coordinated with institutional authorities to ensure implementation.

11.1. Self-Compassionate Mindfulness Psychoeducation Program

1. Psychoeducation Session (Holding Our Own Hand: Discovering Self-Compassion):

   The first session for delinquent adolescents in the experimental group begins with an introduction to the program. Following this, a "Name Ball Game" activity is conducted to facilitate the acquaintance process among group members. The concept of self-compassion is then defined, accompanied by a brief presentation. Participants are introduced to self-compassionate mindfulness practices and meditation techniques, including guidance on how to find a suitable meditation posture. Each participant is provided with a Self-Compassionate Mindfulness Psychoeducation Program booklet, offering them the opportunity to follow the formal and informal practices throughout the process. After completing the practices, participants are invited to share their feedback and suggestions. The session concludes with the assignment of homework. At the end of this session, adolescents are expected to gain an understanding of the concept of self-compassion and learn how to recognize and accept their emotions without self-criticism or blame in the face of challenges.
2. Psychoeducation Session (Discovering Awareness of Thought):

   The second session begins with a warm-up activity titled "Imagine a Picture or Photograph." Following a recap of the previous session, adolescents are encouraged to share their experiences regarding the homework. A definition of mindfulness is provided, and a brief presentation is given on mindfulness and the concept of the "automatic pilot." After engaging in both formal and informal practices, participants offer their feedback and suggestions. The session ends with the assignment of homework. By the end of this session, adolescents are expected to develop an awareness of their emotions and thoughts, recognize the relationship between thoughts and behaviors, and acquire emotion regulation skills by identifying and transforming negative automatic thought patterns. Additionally, the session is designed to help participants become aware of the negative effects of internalized stigma and gain skills to distance themselves from and transform negative self-perceptions.
3. Psychoeducation Session (Understanding Pain, Approaching with Compassion):

   The third session begins with a warm-up activity titled "Perception and Attention." The previous session is summarized, and adolescents are encouraged to share their homework experiences. The concept of painful experiences is introduced, followed by a presentation on the common humanity aspect and the role of self-compassion during painful experiences. After completing formal and informal practices, participants share their thoughts and suggestions. The session ends with a homework assignment. By the end of this session, adolescents are expected to recognize that painful experiences are universal, and that accepting their mistakes and offering themselves compassion contributes to the process of forgiveness. This understanding is anticipated to enhance their capacity to forgive both themselves and others. Additionally, the session aims to help adolescents comprehend the concept of common humanity and realize that pain and struggle are part of being human, thus supporting them in perceiving stigmatizing beliefs not as personal flaws but as part of a shared experience.
4. Psychoeducation Session (Facing Reality: Acceptance):

   The fourth session begins with a warm-up activity titled "Circle of Warm-up." Following a summary of the previous session, adolescents are invited to discuss their experiences with the assigned homework. The concept of self-kindness is defined, and a presentation is provided on acceptance and its significance in self-compassion. After the formal and informal exercises are completed, participants provide feedback and suggestions. The session concludes with a homework assignment. At the end of this session, adolescents are expected to manage stressful moments more effectively and learn to accept negative emotions with less resistance. This is anticipated to enhance their emotion regulation skills and reduce their internal resistance toward forgiving themselves and others, enabling them to see forgiveness as a means of empowerment. Through self-kindness and compassion practices, adolescents are expected to learn how to treat themselves with kindness, reduce self-criticism arising from stigma, and foster a more positive self-view.
5. Psychoeducation Session (Calm Waters: Forgiveness):

   The fifth session begins with a warm-up activity titled "Museum Tour." The session continues with a summary of the previous session and a discussion of participants' homework experiences. The concept of forgiveness is defined, and a presentation on the importance of forgiving oneself and others is delivered. Following the formal and informal exercises, participants provide their feedback and suggestions. The session concludes with a homework assignment. By the end of this session, adolescents are expected to gain the ability to accept and release their past mistakes and negative experiences, helping them to develop a more positive outlook toward themselves and others through the act of forgiveness. Additionally, this session is expected to enhance adolescents' ability to recognize, manage, and cope with negative emotions, thereby fostering the development of emotion regulation skills.
6. Psychoeducation Session (Moving Forward, Farewell, and a New Beginning):

The sixth and final session begins with a warm-up activity titled "Trust Activity." The previous session is reviewed, and participants are invited to share their homework experiences. The entire program is summarized, and a presentation on the application and importance of self-compassion in daily life is delivered. After completing the final formal and informal practices, participants provide feedback on the activities. The session concludes with a comprehensive feedback collection regarding all sessions. By the end of this session, the following outcomes are anticipated for adolescents:

Through meditation, self-compassionate journaling, and mindfulness practices, adolescents are expected to recognize, manage, and express intense and challenging emotions more effectively, thereby developing emotion regulation skills.

Practices related to self-forgiveness, forgiveness of others, and loving-kindness are expected to help adolescents accept their past mistakes and cultivate a more compassionate attitude toward others. As a result, a decrease in negative emotions such as guilt and anger, along with improved forgiveness abilities, is anticipated.

Mindfulness practices focused on self-compassion are expected to enhance adolescents' abilities to cope with negative self-judgments and foster a compassionate and accepting inner voice. This, in turn, is expected to reduce the impact of perceived societal stigma and promote a sense of self-worth and acceptance.

12. Collection of Post-Test Data

One week after the completion of the psychoeducation program sessions applied to the experimental group of juvenile offenders, the "Emotion Regulation Scale for Children and Adolescents," "Forgiveness Scale for Adolescents," and "Internalized Stigma Scale for Children and Adolescents" will be administered to the entire sample group (both experimental and control groups) using the face-to-face interview technique.

13.The statistical evaluation of the data will be carried out by a statistics expert. The data will be analyzed using the IBM SPSS V23 software. In the statistical evaluation of the data in the study, the following tests will be used:

Skewness and kurtosis coefficients to determine the conformity of the data to normal distribution,

Frequency and percentage distribution to determine the descriptive characteristics of the adolescents in the experimental and control groups,

Chi-square test (Pearson chi-square test, Fisher-Freeman-Halton test, Fisher's Exact test) and Independent Samples t-test to compare the descriptive characteristics of the adolescents in the experimental and control groups,

Independent Samples t-test to compare the pre-test and post-test values of the adolescents in the experimental and control groups,

Two-factor ANOVA for mixed measurements (Pillai's Trace Test) to compare the changes observed in two different measurements in terms of total/subscale scores of the scales according to the experimental and control groups,

If necessary, Missing Completely at Random (MCAR) analysis will be used for missing data,

Cronbach's Alpha Reliability Coefficient will be used to determine the internal consistency coefficients of the total/subscale scores of the scales.

14. Ethical Considerations Approval for the study was obtained from the Ethics Committee for Social and Human Sciences Research at Ondokuz Mayıs University . Based on this approval, institutional permission was granted by the Ministry of Justice for the study to be conducted at the Kavak Juvenile and Youth Closed Penal Institution in Samsun . The researcher holds the necessary certifications related to "Self-Compassionate Mindfulness" . Permissions for the use of the "Emotion Regulation Scale for Children and Adolescents," the "Forgiveness Scale for Adolescents," and the "Internalized Stigma Scale for Children and Adolescents" were obtained from the scale developers via email . Informed consent forms were obtained both verbally and in writing from the adolescents included in the study. Confidentiality of the data was maintained by the research team throughout the entire study process.

ELIGIBILITY:
Inclusion Criteria:

* Being literate

Being able to speak and understand Turkish

Being between 12 and 18 years of age

Having been convicted and currently incarcerated

Willingness to participate in the study

Exclusion Criteria:

* Unwillingness to participate in the study

Having a psychiatric diagnosis that may disrupt group dynamics

Being younger than 12 or older than 18 years of age

Having a physical disability that may affect participation in the study (e.g., hearing, speech impairments, etc.)

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Forgiveness Scale for Adolescents | From enrollment until the end of the 6-week psychoeducation program
  The Forgiveness Scale for Adolescents (FSA), developed by Asıcı and Karaca (2018), is a 21-item, 5-point Likert-type scale (1 = Does not describe me at all, 5 = Describes me completely) designed to measure adolescents' tendency to forgive in interpersonal relationships. The FSA includes four subscales that reflect components of forgiveness: revenge, holding a grudge, and empathy.
  Higher scores on each subscale indicate a stronger presence of the trait measured by that subscale. In addition, a total score can be obtained from the scale. Total scores range from 21 to 105, with higher scores indicating a higher tendency to forgive. In this study, only the total scores from the scale were used.
  In the scale development study, the Cronbach's alpha coefficient for the entire scale was calculated as .90, indicating high internal consistency.
Emotion Regulation Scale for Children and Adolescents | From enrollment until the end of the 6-week psychoeducation program
  The scale was developed by Phillips and Power (2007) and its validity and reliability study was conducted by Yıldız and Duy (2014). The scale consists of 18 items and is scored on a 5-point Likert scale. It includes four sub-dimensions: Internal Functional Emotion Regulation (IFER), External Functional Emotion Regulation (EFER), Internal Dysfunctional Emotion Regulation (IDER), and External Dysfunctional Emotion Regulation (EDER). As the scores on the sub-dimensions increase, it indicates that the adolescent more frequently uses the emotion regulation strategy represented by that sub-dimension. Conversely, lower scores suggest less frequent use of that strategy.
  According to Yıldız and Duy (2014), the test-retest reliability coefficients obtained by administering the scale to 175 students with a two-week interval were reported as follows: 0.51 for the internal functional emotion regulation sub-dimension, 0.70 for the external dysfunctional emotion regulation sub-dimension, 0.56 for t
Internalized Stigma Scale for Children and Adolescents | From enrollment until the end of the 6-week psychoeducation program
  The Internalized Stigma Scale for Children and Adolescents was developed by Çağlayan (2019). The scale consists of 32 items grouped under six factors:
  Behavioral Problems (25 items): Children and adolescents with emotional and behavioral problems often get into fights.
  Social and Academic Adjustment (8 items): Children and adolescents with emotional and behavioral problems are considered unreliable.
  Concealment of Diagnosis (3 items): Individuals with emotional and behavioral problems make an effort to keep their issues a secret.
  Feelings of Exclusion (1 item): Children and adolescents with emotional and behavioral problems engage in self-harming behaviors.
  Chronicity of the Problem (5 items): Individuals with emotional and behavioral problems feel bad because of their diagnosis.
  Emotional Difficulties (19 items): Children and adolescents with emotional and behavioral problems often feel lonely.
  The total score that can be obtained from the scale ranges between 32 and 160.

IPD SHARING:
Plan to Share IPD: No